CLINICAL TRIAL: NCT02931916
Title: Evaluation of Reliability and Validity of a Smart-phone Application Designed for Chronic Ankle Instability Subjects' Postural Control Assessment
Brief Title: Evaluation of Reliability and Validity of a Smart-phone Postural Control Assessment Application
Status: Completed | Type: Observational
Sponsor: National Yang Ming Chiao Tung University (Other)
Collaborators: Ministry of Science and Technology, Taiwan (Other Government)
Responsible Party: Principal Investigator, Wen-Hsu Sung, professor, National Yang Ming Chiao Tung University
Other Study IDs: 2016CAIAppR&V
Record Dates: First submitted 2016-09-29; First posted 2016-10-13 (Estimated); Last update posted 2018-10-25 (Actual); Status verified 2018-10

CONDITIONS: Other Instability, Ankle and Foot
Keywords: smart-phone; assessment; chronic ankle instability

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- healthy group: recruited for evaluation of system reliability
- Chronic Ankle Instability group: recruited for evaluation of system validity

SUMMARY:
The purpose of this study is to evaluate the reliability and validity of smart-phone based system in postural control ability assessment on subjects with chronic ankle instability.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of ankle functional instability

Exclusion Criteria:

* any other condition would affect postural control performance

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: chronic ankle instability group
Sampling Method: Probability Sample
Enrollment: 138 (Actual)
Dates: Start 2016-11; Primary Completion 2018-03-30 (Actual); Study Completion 2018-08-31 (Actual)

PRIMARY OUTCOMES:
physiological parameter: acceleration data from built-in sensor with unit: m/s^2 | 40 seconds
  Using the built-in sensor to record the acceleration data during each seconds trial.
  Both x, y and z axialis will be recorded
physiological parameter: orientation data from built-in sensor with unit: degree | 40 seconds
  Using the built-in sensor to record the acceleration data during each seconds trials.
  Both x, y and z axialis will be recorded

CONTACTS AND LOCATIONS:
Locations (1):
- Yang Ming university, Taipei, Taiwan